CLINICAL TRIAL: NCT06206837
Title: AN INTERVENTIONAL SAFETY AND EFFICACY PHASE 1B/2, OPEN-LABEL STUDY TO INVESTIGATE TOLERABILITY, PK, AND ANTITUMOR ACTIVITY OF VEPDEGESTRANT (ARV-471/PF-07850327), AN ORAL PROTEOLYSIS TARGETING CHIMERA, IN COMBINATION WITH PF-07220060 IN PARTICIPANTS AGED 18 YEARS AND OLDER WITH ER+/HER2- ADVANCED OR METASTATIC BREAST CANCER
Brief Title: A Study to Learn About Vepdegestrant When Given With PF-07220060 to People With Advanced or Metastatic Breast Cancer.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4891026; TACTIVE-K (Other: Alias Study Number); 2023-508130-33-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-12-13; First posted 2024-01-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Proteolysis Targeting Chimera (PROTAC); metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1b will use an escalation/de-escalation approach to determine the recommended phase 2 dose (RP2D) of vepdegestrant when administered in combination with PF-07220060. The decision to escalate the starting dose level of vepdegestrant will be using mTPI-2 decision criteria based on the number of dose limiting toxicity (DLT)-evaluable participants and the number of DLTs in those participants during the DLT observation period (Cycle 1).
  Phase 2 will further evaluate the preliminary antitumor activity and safety of the combination RP2D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- vepdegestrant in combination with PF-07220060 (Experimental): vepdegestrant administered orally once daily (QD) continuously and PF-07220060 administered orally twice daily (BID) continuously on 28-day cycles
  Interventions: Drug: vepdegestrant; Drug: PF-07220060

INTERVENTIONS:
Drug: vepdegestrant — Daily oral dosages of vepdegestrant continuously, dose escalation/de-escalation in Phase 1b until recommended phase 2 dose (RP2D) determined, cycles lasting 28 days
  Other Names: ARV-471 / PF07850327
Drug: PF-07220060 — Daily oral dosages of PF-07220060 continuously, dose escalation/de-escalation in Phase 1b until recommended phase 2 dose (RP2D) determined, cycles lasting 28 days

SUMMARY:
The purpose of this study is to learn about the safety and effects of giving vepdegestrant along with PF-07220060. Vepdegestrant is studied to see if it can be a possible treatment for advanced metastatic breast cancer. This type of cancer would have spread from where it started (breast) to other parts of the body and would be tough to treat. The study is seeking for participants who have breast cancer that:

* is hard to treat (advanced) and may have spread to other organs (metastatic).
* is sensitive to hormonal therapy (it is called estrogen receptor positive).
* is no longer responding to treatments taken before starting this study.

All the participants will receive vepdegestrant and PF-07220060. Both medicines will be taken by mouth. The medicines will be taken at home. The experience of people receiving the study medicines will be studied. This will help see if the study medicines are safe and effective. Participants will continue to take vepdegestrant and PF-07220060 until:

* their cancer is no longer responding, or
* side effects become too severe. They will have visits at the study clinic about every 4 weeks.

DETAILED DESCRIPTION:
C4891026 is a prospective, open-label, multicenter, Phase 1b/2 study to evaluate the safety, antitumor activity, and pharmacokinetic (PK) of vepdegestrant in combination with PF-07220060 in the treatment of participants with Estrogen Receptor Positive/Human Epidermal Growth Factor Receptor 2 Negative (ER+/HER2-) Advanced or Metastatic Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of breast cancer. At time of enrollment this must not be amenable to surgical resection with curative intent (≥1% ER+ stained cells as per local practice on the most recent tumor biopsy HER2- tumor by IHC or in-situ hybridization per ASCO/CAP).
* prior anticancer therapies: Phase 1b: at least 1 line of SOC for A/MBC; Prior fulvestrant allowed; ≤1 prior chemotherapy line (no antibody-drug conjugates permitted) for A/MBC setting allowed. Phase 2: At least one and maximum 2 lines of ET in A/MBC setting and most recent ET-based regimen for >6 months.

  1, and only 1, prior CDK4/6 inhibitor-based regimen required. Up to 1 prior regimen of cytotoxic chemotherapy (no antibody-drug conjugates permitted) in the A/MBC setting; Prior fulvestrant allowed.
* Participant with only non-measurable lesion (Phase1b) or at least 1 measurable lesion as defined by RECIST v1.1. (Phase2) are eligible.
* ECOG PS = 0 or 1 (Phase1b) ; ≤2 (Phase2)

Exclusion Criteria:

* visceral crisis at risk of life-threatening complications in the short term.
* Any condition precluding an adeguate absorption of study interventions.
* newly diagnosed brain metastases, or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease. Participants with a history of CNS metastases or cord compression are eligible if they have been definitively treated, clinically stable and discontinued anti-seizure medications and corticosteroids for at least 28 days prior to enrollment in the of study.
* history of any other tumor malignancies within the past 3 years, except for the following: (1) adequately treated basal or squamous cell carcinoma of the skin; (2) curatively treated in situ carcinoma of the cervix. Inflammatory breast cancer are excluded
* impaired cardiovascular function or clinically significant cardiovascular diseases.
* concurrent administration of medications, food, or herb supplements that are strong inhibitors/inducers of CYP3A or UGT2B7, moderate inducers of CYP34 (Phase1b only) and drugs known to predispose to Torsade de Pointes or QT interval prolongation.
* renal impairment, not adequate liver function and/or bone marrow function.
* known active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Number of Participants With Dose Limiting Toxicities | 28 days
  Dose Limiting Toxicities (DLTs) rate for Vepdegestrant in combination with PF-07220060, estimated based on data from DLT-evaluable participants during the DLT observation period (Cycle 1).
Phase 2: Percentage of Participants With Objective Response by investigator assessment | Up to approximately 1 year
  Objective response (OR) refers to confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1. as determined by investigator assessment.

SECONDARY OUTCOMES:
Phase 1b and Phase 2: Evaluation of Safety of Vepdegestrant in combination with PF-07220060 (number of participants experiencing any AE, SAE, treatment-related AE and treatment-related SAE) | First study drug dose through a minimum of 28 Days After Last study drug administration
  An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. A severe adverse event (SAE) is any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect and other important medical events. A treatment-related AE is any untoward medical occurrence attributed to study drug in a participant who received study drug.
  AEs were graded by the investigator according to the CTCAE version 5.0 and coded using MedDRA were reported. Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening or disabling; and Grade 5=death.
Phase 1b and Phase 2: Evaluation of Safety of Vepdegestrant in combination with PF-07220060 (number of participants with lab abnormalities - Hematology and coagulation parameters) | First study drug dose through a minimum of 28 Days After Last study drug administration
  Blood samples were collected for the analysis of the following hematology and coagulation parameters: hemoglobin [g/L], platelets, leukocytes, neutrophils, lymphocytes, monocytes, eosinophils and basophils [10^9/L]; partial thromboplastin time prolonged and prothrombin time [seconds]; international normalized ratio increased. Number of participants with hematological and coagulation abnormalities by grade as per Common Terminology Criteria for Adverse Events (CTCAE version 5.0) were reported. Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening or disabling; and Grade 5=death. For laboratory tests without CTCAE grade definitions, results will be categorized as normal, abnormal, or not done.
Phase 1b and Phase 2: Evaluation of Safety of Vepdegestrant in combination with PF-07220060 (number of participants with lab abnormalities - chemistry parameters) | First study drug dose through a minimum of 28 Days After Last study drug administration
  Blood samples were collected for analysis of clinical chemistry parameters. These included: alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, [international unit per liter (IU/L)] ; Lipase and amilase [IU/L] (limited to cycle1 only); Albumin, bilirubin, urea ,calcium, creatinine, glucose, magnesium, phosphate, uric acid chloride, potassium and sodium [millimol per liter (mmol/L)]; eGFR [milliliter per minute (ml/min)]. Number of participants with hematological and coagulation abnormalities by grade as per Common Terminology Criteria for Adverse Events (CTCAE version 5.0) were reported. Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening or disabling; Grade 5=death. For laboratory tests without CTCAE grade definitions, results will be categorized as normal, abnormal, or not done.
Phase 1b and Phase 2: Evaluation of Safety of Vepdegestrant in combination with PF-07220060 (number of participants with changes from baseline for ECG parameters) | First study drug dose through a minimum of 28 Days After Last study drug administration
  The following ECG parameters were analyzed and changes from baseline were assessed : heart rate, PR interval, QT interval, QRS interval and QT interval corrected using Fridericia's formula (QTcF).
Phase 1b and Phase 2: Evaluation of Tolerability of Vepdegestrant in combination with PF-07220060 (number of participants experiencing any AE, SAE, treatment-related AE and treatment-related SAE) | First study drug dose through a minimum of 28 Days After Last study drug administration
  "An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. A severe adverse event (SAE) is any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect and other important medical events. A treatment-related AE is any untoward medical occurrence attributed to study drug in a participant who received study drug.
  AEs were graded by the investigator according to the CTCAE version 5.0 and coded using MedDRA where reported. Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening or disabling; and Grade 5=death."
Phase 1b and Phase 2: Evaluation of Tolerability of Vepdegestrant in combination with PF-07220060 (number of participants with lab abnormalities- Hematology and coagulation parameters) | First study drug dose through a minimum of 28 Days After Last study drug administration
  Blood samples were collected for the analysis of following hematology and coagulation parameters: hemoglobin [g/L], platelets, leukocytes, neutrophils, lymphocytes, monocytes, eosinophils and basophils [10^9/L]; partial thromboplastin time prolonged and prothrombin time [seconds]; international normalized ratio increased. Number of participants with hematological and coagulation abnormalities by grade as per Common Terminology Criteria for Adverse Events (CTCAE version 5.0) were reported. Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening or disabling; and Grade 5=death. For laboratory tests without CTCAE grade definitions, results will be categorized as normal, abnormal, or not done.
Phase 1b and Phase 2: Evaluation of Tolerability of Vepdegestrant in combination with PF-07220060 (number of participants with lab abnormalities - chemistry parameters) | First study drug dose through a minimum of 28 Days After Last study drug administration
  Blood samples were collected for analysis of clinical chemistry parameters. These included: alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, [international unit per liter (IU/L)] ; Lipase and amilase [IU/L] (limited to cycle1 only); Albumin, bilirubin, urea ,calcium, creatinine, glucose, magnesium, phosphate, uric acid chloride, potassium and sodium [millimol per liter (mmol/L)]; eGFR [milliliter per minute (ml/min)]. Number of participants with hematological and coagulation abnormalities by grade as per Common Terminology Criteria for Adverse Events (CTCAE version 5.0) were reported. Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening or disabling; and Grade 5=death. For laboratory tests without CTCAE grade definitions, results will be categorized as normal, abnormal, or not done.
Phase 1b and Phase 2: Evaluation of Tolerability of Vepdegestrant in combination with PF-07220060 (number of participants with changes from baseline for ECG parameters) | First study drug dose through a minimum of 28 Days After Last study drug administration
  Following ECG parameters were analyzed and changes from baseline were assessed: heart rate , PR interval, QT interval, QRS interval and QT interval corrected using Fridericia's formula (QTcF).
Phase 1b: To evaluate antitumor activity of Vepdegestrant in combination with PF-07220060 | Up to approximately 1 year
  Objective response (OR) refers to confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1. as determined by investigator assessment.
Phase 1b and Phase 2: Duration of Response by investigator assessment. | Up to approximately 1 year
  Duration of Response (DoR) is defined for participants with confirmed OR (CR or PR) as the time from the first documentation of OR to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Phase 1b and Phase2: Percentage of participants with Clinical Benefit Response by investigator assessment. | Up to approximately 1 year
  Clinical Benefit Response (CBR) is defined as the proportion of participants with Best Overall Response of confirmed CR or PR at any time, or Stable Disease (SD) ≥24 weeks
Phase 1b and Phase 2: Progression Free Survival by investigator assessment. | Up to approximately 1 year
  Progression Free Survival (PFS) is defined as the time from the date of first dose of study interventions to the date of first documentation of PD or death due to any cause, whichever occurs first.
Phase 1b and Phase 2: Plasma concentrations of Vepdegestrant, ARV-473 and PF-07220060 when given in combination. | Phase 1b: Pre-dose Day 8; Pre-, 0.5, 1, 2, 4, 6, 8, 12h post-dose Day 15; Pre- and 4-8h post-dose 29; Pre- and 4-8h post-dose Day 43; Pre-dose Days 57, 113 and 169. Phase 2: Pre- and 4-8h post-dose Days 15, 29 and 43; Pre-dose Days 57, 113 and 169
  To evaluate the plasma exposure of vepdegestrant, ARV-473, and PF-07220060 when vepdegestrant and PF-07220060 are given in combination.
Phase 1b: Evaluation of the PK of Vepdegestrant and PF-07220060 when given in combination | Phase 1b (a cycle is 28 days): Pre-dose on Day 8 of Cycle 1; Pre-dose, 0.5, 1, 2, 4, 6, 8, 12h post-dose on Day 15 of Cycle 1; Pre-dose and 4-8h on Day 1 of Cycle 2; Pre-dose and 4-8h post-dose on Day 15 of Cycle 2; Pre-dose on Day 1 of Cycles 3, 5 and 7
  Steady-state Cmax (maximum observed serum concentration of drug [Micrograms per milliliter]) of vepdegestrant, ARV-473, and PF-07220060.
Phase 1b: Evaluation of the PK of Vepdegestrant and PF-07220060 when given in combination | Phase 1b (a cycle is 28 days): Pre-dose on Day 8 of Cycle 1; Pre-dose, 0.5, 1, 2, 4, 6, 8, 12h post-dose on Day 15 of Cycle 1; Pre-dose and 4-8h on Day 1 of Cycle 2; Pre-dose and 4-8h post-dose on Day 15 of Cycle 2; Pre-dose on Day 1 of Cycles 3, 5 and 7
  Steady-state Tmax (time taken (in hours) to reach the maximum serum drug concentration) of vepdegestrant, ARV-473, and PF-07220060.
Phase 1b: Evaluation of the PK of Vepdegestrant and PF-07220060 when given in combination | Phase 1b (a cycle is 28 days): Pre-dose on Day 8 of Cycle 1; Pre-dose, 0.5, 1, 2, 4, 6, 8, 12h post-dose on Day 15 of Cycle 1; Pre-dose and 4-8h on Day 1 of Cycle 2; Pre-dose and 4-8h post-dose on Day 15 of Cycle 2; Pre-dose on Day 1 of Cycles 3, 5 and 7
  Steady-state AUClast (Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) of vepdegestrant, ARV-473, and PF-07220060.
Phase 2:ctDNA plasma quantitative changes from pre-treatment | Phase 2 (each cycle is 28 days): Pre-dose on Day 1 of Cycles 1, 2 and 3 and after last treatment administration.
  To assess changes from baseline levels in plasma circulating tumor DNA (ctDNA) with treatment and to evaluate potential predictability of their associations with clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- United States (30):
  - Highlands Oncology, Fayetteville, Arkansas
  - Highlands Oncology, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Hoag Health Center Irvine, Irvine, California
  - Hoag Hospital Irvine, Irvine, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford Cancer Center, Palo Alto, California
  - Stanford Cancer Institute - Clinical Trials Office, Palo Alto, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - UCHealth Poudre Valley Hospital, Fort Collins, Colorado
  - UCHealth Harmony, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth - Medical Center of the Rockies, Loveland, Colorado
  - Smilow Cancer Hospital - Yale New Haven Health, New Haven, Connecticut
  - Yale - New Haven Hospital - Yale Cancer Center, New Haven, Connecticut
  - Smilow Cancer Hospital Phase 1 Unit, New Haven, Connecticut
  - Smilow Cancer Hospital - Trumbull, Trumbull, Connecticut
  - START Midwest, Grand Rapids, Michigan
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack, Commack, New York
  - MSK Westchester, Harrison, New York
  - Rockefeller Outpatient Pavilion (53rd Street), New York, New York
  - Evelyn H. Lauder Breast and Imaging Center (BAIC)., New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MSK Nassau, Uniondale, New York
  - START San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - START Mountain Region, West Valley City, Utah
- Belgium (4):
  - Antwerp University Hospital, Edegem, Antwerpen
  - Institut Jules Bordet, Anderlecht, Bruxelles-capitale, Région de
  - UZ Leuven, Leuven, Vlaams-brabant
  - AZ Groeninge Campus Kennedylaan, Kortrijk, West-vlaanderen
- Canada (3):
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Wuhan Union Hospital Cancer Center, Wuhan, Hubei
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
- France (3):
  - Institut Régional du Cancer Montpellier, Montpellier, Hérault
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire-atlantique
  - Institut Paoli-Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
- Japan (4):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kanagawa cancer center, Yokohama, Kanagawa
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Showa Medical University Hospital, Tokyo
- Puerto Rico (3):
  - BRCR Global - Mayaguez Administrative Office, Mayagüez
  - BRCR Global - Mayagüez, Mayagüez
  - Pan American Center for Oncology Trials, LLC, Rio Piedras
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida, Lleida [lérida]
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891026